CLINICAL TRIAL: NCT03820934
Title: A Prospective, Validation Study of FibroSURE™ and FibroScan® as Screening, Detection, and Monitoring Alternatives to Liver Biopsy for Methotrexate-induced Hepatic Fibrosis and Cirrhosis in Patients With Psoriasis
Brief Title: FibroScan ® Study: Assessing Liver Fibrosis in Patients Using Methotrexate for Psoriasis
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Per Investigator study was terminated prematurely
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Principal Investigator, Neil Korman, Director, Clinical Trials Unit, University Hospitals Cleveland Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 12-17-09
Record Dates: First submitted 2019-01-15; First posted 2019-01-29 (Actual); Last update posted 2020-07-23 (Actual); Status verified 2020-07

CONDITIONS: Psoriasis
Keywords: Methotrexate; FibroScan; FibroSure; Cirrhosis; Fibrosis
MeSH Terms: conditions — Psoriasis; Fibrosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Patients undergoing Fibroscan and Fibrosure (Other): Patient's will undergo fibroscan and fibrosure to test their liver for the level of liver fibrosis as measured by these test. The scores from these tests will then be compared to the amount of fibrosis noted on a standard of care liver biopsy.
  Interventions: Diagnostic Test: Fibroscan and Fibrosure

INTERVENTIONS:
Diagnostic Test: Fibroscan and Fibrosure — Patient's will undergo fibroscan and fibrosure to test their liver for the level of liver fibrosis as measured by these tests. Fibroscan uses vibrations sent through the liver to measure its stiffness and the fibrosure uses laboratory and demographic parameters to create a score associated with a certain level of fibrosis. The scores from these tests will then be compared to the amount of fibrosis noted on a standard of care liver biopsy.

SUMMARY:
The purpose of this study is to validate FibroScan and FibroSURE™ as equal or superior alternatives to liver biopsy for the monitoring and detection of methotrexate-induced hepatic fibrosis and cirrhosis in patients with moderate-to-severe psoriasis.

DETAILED DESCRIPTION:
The goals of this study are to validate FibroScan and FibroSURE™ as equal or superior alternatives to liver biopsy. The goal is to evaluate the monitoring and detection of methotrexate-induced hepatic fibrosis and cirrhosis in patients with moderate-to-severe psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* Male or female greater than or equal to 18 years of age
* Must have a diagnosis of moderate-to-severe psoriasis
* Newly starting methotrexate

Exclusion Criteria:

* Allergy to methotrexate
* History of chronic alcohol abuse
* Diagnosis of liver disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-02-10 (Actual); Primary Completion 2019-05-15 (Actual); Study Completion 2019-05-15 (Actual)

PRIMARY OUTCOMES:
Fibrosis Score Correlation | 5 years
  The correlation between the clinical fibrosis scores generated by the FibroScan® and FibroSURE™ alone and in combination to the METAVIR fibrosis score generated from the histologic review of a liver biopsy performed for the assessment of liver fibrosis in a psoriasis patient who reaches a cumulative methotrexate dose of 1g.

SECONDARY OUTCOMES:
Fibrosis Score Validity to Liver Biopsy Results | 5 years
  Determine if the clinical fibrosis scores generated by the FibroScan® and FibroSURE™ alone and in combination can be safely used as alternatives to performing a liver biopsy when screening for liver fibrosis in psoriasis patients who have reached a cumulative methotrexate dose of 1 gram

CONTACTS AND LOCATIONS:
Overall Officials: Neil Korman, MD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals Cleveland Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided